CLINICAL TRIAL: NCT05483764
Title: Ultrasonographic Measurements of the Achilles Tendon and Talar Condylar Cartilage Thickness in Paraplegia Patients.
Status: Active, not recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-SK-03
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Paraplegia
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paraplegia
  Interventions: Device: Ultrasonographic evaluations
- Control
  Interventions: Device: Ultrasonographic evaluations

INTERVENTIONS:
Device: Ultrasonographic evaluations — Ultrasonographic evaluations of the talar cartilage will be performed with an 8 MHz linear probe (B-K Medical Ultrasound Scanner Class I Type B) by the same physiatrist according to the European Musculoskeletal Ultrasound Study Group (EURO-MUSCULUS).
  Ultrasonographic evaluations of the Achilles tendon will be performed by the same physiatrist with an 8 MHz linear probe (B-K Medical Ultrasound Scanner Class I Type B) according to the European Musculoskeletal Ultrasound Study Group (EURO-MUSCULUS).

SUMMARY:
Investigators aim to measure the ankle talar cartilage and achilles tendon thicknesses ultrasonographically in paraplegic patients and compare them with the normal population.

DETAILED DESCRIPTION:
Paraplegia is a clinical condition that expresses the loss of motor and sensory function in the lower extremities after spinal cord injury. A specialized and intensive rehabilitation program is needed in these patient groups who develop immobilization. In healthy individuals, there is a certain biomechanics of the lower extremity. In paraplegic patients, this biomechanics changes due to weakness in the lower extremities. These biomechanical changes can cause different loads and effects on the lower extremity joints, muscles, tendons, and articular cartilages of paraplegic patients. Among the rehabilitation goals of paraplegic patients, it is to stand up and walk the patient with or without support, with or without a device. During this rehabilitation, the position and function of the ankle is important. In this process, the talar condylar cartilage and achilles tendon forming the ankle joint can be exposed to different loads.

Ultrasonography is frequently used in physical therapy practice because it does not contain any radiation, has no side effects to the patient, facilitates dynamic and real-time evaluation of joint and muscle conditions and functions, and provides guidance during interventional procedure planning. In this study, investigators aim to ultrasonographically measure ankle talar cartilage and Achilles tendon thicknesses in paraplegic patients with long-term immobilization and compare them with the normal population.

Our study will be organized as a observational study. It is planned to include 20 paraplegia patients and 20 healthy volunteers in the study.

Demographic data of the patients and healthy volunteers will be recorded. Paraplegia patients will be evaluated in terms of Barthel Index, Modified Ashworth Scale, American Spinal Injury Association (ASIA) scale, Walking Index for Spinal Cord Injury Scale (WISCII-2).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are paraplegic after traumatic spinal cord injury (ASIA A-D)
* Healthy volunteers older than 18 years for control patients.

Exclusion Criteria:

* Patients who had a previous trauma-related operation on the ankle.
* Patients who had fixed contracture or severe spasticity on the ankle.
* Patients who had lower-limb length difference of more than 2 cm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group will be composed of healthy individuals who are compatible with the patient group in terms of age, gender and weight.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Ankle talar cartilage thicknesses | 1 day
  Patients will lie on the examination table supine with their knees flexed to 90 degrees and ankles in a flat-footed position. The probe was placed mid-longitudinally over the ankle joint to assess the cartilage of the talar dome. The articular cartilage will be displayed as an anechoic line between bony cortex and adipose tissue. Cartilage thickness will be measured by drawing a straight line from the bone-cartilage interface to the cartilage-fatty tissue interface at the midpoint of the talar dome. The thickness of the hyaline cartilage will be measured in centimeters (cm).
Achilles tendon thicknesses | 1 day
  Ultrasound (US) evaluation will be performed with patients in the prone position on examination table with their feet in 90 degrees of flexion. Achilles tendon of the each patient and healthy volunteer will be scanned.
  Antero-posterior achilles thickness will be measured on the same mid-longitudinally scan at two different levels: at the insertion of the achilles tendon deeper edge into the calcaneal bone and 3 cm more proximal. The thickness of the achilles tendon will be measured in centimeters (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)